CLINICAL TRIAL: NCT07050342
Title: Evaluation Der Spezialambulanz Ernährung Und Psyche: Eine Pilotstudie
Brief Title: Evaluation of the Specialized Clinic for Nutrition and Mental Health: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1300/2024
Record Dates: First submitted 2025-05-06; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Psychosomatic Disorders; Mental Health Care
Keywords: Nutritional Psychiatry; Psychosomatic Disorders; Stress Reduction; Personalized Nutrition; Mental Health
MeSH Terms: conditions — Psychophysiologic Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition-Based Psychosomatic Care (Experimental): Participants receive individualized, nutrition-focused care as part of standard treatment in a psychosomatic outpatient clinic. The study observes changes in stress levels, psychological well-being, quality of life, and relevant blood biomarkers over 12 months. No experimental treatment is administered. Participants complete questionnaires and undergo routine blood tests every 3 months.
  Interventions: Other: Personalized Nutrition-Based Psychosomatic Care

INTERVENTIONS:
Other: Personalized Nutrition-Based Psychosomatic Care — This intervention involves personalized, nutrition-focused care provided in a specialized outpatient clinic for individuals with psychosomatic and mental health conditions. The care model integrates nutritional counseling, education on gut-brain interactions, and patient-centered support to promote psychological well-being and reduce stress. No experimental drugs or diets are administered. Instead, the intervention focuses on individualized recommendations based on clinical assessments and ongoing routine laboratory markers (e.g., inflammatory markers, vitamin levels). Participants also receive guidance aimed at improving dietary habits and resilience within a biopsychosocial framework. The intervention is part of regular clinical care and not blinded or randomized.
  Other Names: Nutritional Psychiatry Intervention

SUMMARY:
The goal of this observational pilot study is to learn how personalized nutrition-focused care can help people with mental and psychosomatic health problems. This study takes place in Europe's first outpatient clinic that focuses on how diet affects mental well-being.

The main questions the study aims to answer are:

Does care at this clinic help lower participants' stress levels over one year?

Do participants report better mental health, resilience, and quality of life during the study?

Are improvements in mental health linked to changes in diet and blood markers like inflammation?

Participants will:

Fill out online questionnaires every 3 months over one year. These ask about stress, physical symptoms, quality of life, diet, and satisfaction with care.

Give small blood samples during their regular clinic visits. These samples will be checked for common health markers such as inflammation.

This study will help researchers understand whether nutrition-focused care can support mental and physical health, and whether this approach should be tested in larger future studies.

DETAILED DESCRIPTION:
Detailed Description

This is a prospective, monocentric pilot study evaluating the effectiveness of a novel, personalized, nutrition-based outpatient care model for individuals with mental and psychosomatic disorders. The study is conducted at the Department of Medical Psychology, Psychosomatics, and Psychotherapy at the Medical University of Graz, Austria. It is the first clinical research initiative to systematically evaluate outcomes of care at Europe's first outpatient clinic specializing in the relationship between diet and mental health, operating under the framework of Nutritional Psychiatry and Nutritional Psychosomatics.

Background and Rationale Psychiatric and psychosomatic disorders are among the most prevalent and disabling health conditions globally. Conventional treatments-primarily pharmacotherapy and psychotherapy-are often insufficient. Approximately 20-30% of patients remain treatment-resistant despite intensive interventions, suffering from persistent symptoms such as fatigue, pain, sleep disturbances, and cognitive impairments. Additionally, rising incidence rates further highlight the need for innovative, integrative approaches.

Nutritional Psychiatry, a rapidly growing field, examines how dietary patterns and nutritional status impact mood, stress response, and physical symptoms, particularly through mechanisms such as the gut-brain axis. Disruptions in the gut microbiome, linked to poor dietary quality, have been shown to increase systemic inflammation and dysregulate neurotransmitter metabolism, such as serotonin. Research suggests that dietary interventions-especially anti-inflammatory diets rich in omega-3 fatty acids, fiber, and antioxidants (e.g., Mediterranean diet)-can contribute to mental well-being and may play a supportive role in psychosomatic treatment.

The outpatient clinic for Nutrition and Psychosomatics at the LKH Graz offers individualized care incorporating personalized dietary counseling and education, lifestyle guidance, and psychosocial support. The approach is grounded in a salutogenetic model, focusing not only on symptom reduction but also on strengthening health resources and resilience.

Objectives and Hypotheses This pilot study aims to collect preliminary data on the effectiveness of the clinic's integrative care model, focusing on changes in self-reported stress and psychological well-being over a 12-month period. It also seeks to explore potential associations between psychosocial outcomes and physiological parameters such as inflammatory markers.

Primary objective:

To determine whether there is a statistically significant reduction in perceived stress (measured via the Perceived Stress Scale, PSS-10) after one year of care in the outpatient clinic.

Primary hypothesis (H1):

There will be a statistically significant reduction in perceived stress after 12 months of care.

Null hypothesis (H0):

There will be no statistically significant change in perceived stress over the same period.

Secondary objectives include:

Assessing changes in resilience, quality of life, and somatic symptoms.

Evaluating patient satisfaction and subjective health literacy.

Monitoring changes in dietary habits and blood-based biomarkers.

Study Design and Setting This is a non-randomized, single-center, longitudinal, prospective pilot study with repeated measures. Participants will be followed for 12 months, with data collection occurring at baseline and every 3 months thereafter.

Participants are referred by psychiatrists or general practitioners and recruited during their first visit at the clinic. Eligibility screening, informed consent, and baseline assessment occur as part of routine intake procedures. Participation is voluntary, and consent must be provided in writing.

Assessments and Data Collection Self-report instruments will be administered digitally via the EvaSys platform. Participants receive email invitations with secure links to complete the questionnaires online at baseline and every 3 months.

Psychological and health questionnaires include:

Perceived Stress Scale (PSS-10)

Short Form Health Survey (SF-12)

Brief Resilience Scale (BRS-D)

Somatic Symptom Scale (SSS)

EQ-5D-5L

Patient satisfaction questionnaire (adapted from other LKH outpatient services)

NutriMental Screener (baseline only)

Food Frequency Items (baseline and follow-up)

Health literacy is assessed by both patients and their treating physicians using a 10-point Likert scale.

Clinical and demographic variables include: age, sex, BMI, chronic illnesses, psychiatric diagnosis, current medication, smoking status, education, and employment status.

Blood samples are collected as part of routine clinical follow-up at the clinic every 3 months (i.e., not solely for research purposes). Approximately 45 mL of blood will be drawn and analyzed for:

Differential blood count

C-reactive protein (CRP)

Interleukin-6 (IL-6)

Fasting glucose, HOMA-Index

Lipid profile (total cholesterol, HDL, LDL, triglycerides)

Liver enzymes (ALT, AST, GGT)

Kidney function (creatinine, urea)

Electrolytes, uric acid

Vitamin D, vitamin B12, ferritin, homocysteine

No experimental treatment or study-specific intervention will be administered.

Sample Size and Statistical Analysis As a pilot study, no formal sample size calculation was performed. Based on clinic records (Jan-Aug 2024: 91 new patients), approximately 10 new patients are expected per month. Assuming a 70% participation rate, the projected sample size is ~84 participants over 12 months.

Quantitative data will be analyzed using IBM SPSS. Descriptive statistics will summarize baseline characteristics. Changes over time will be examined using paired t-tests and repeated-measures ANOVA. Normality assumptions will be assessed using the Shapiro-Wilk or Kolmogorov-Smirnov test.

Correlational analyses (Pearson or Spearman, depending on data distribution) will examine associations between psychological variables and biological markers. Significance is set at p < 0.05. Qualitative feedback from open-ended survey responses will be analyzed thematically to capture common themes related to patient experience.

Ethical and Legal Considerations This study complies with the Declaration of Helsinki and all relevant national and institutional regulations. Ethics approval has been obtained from the responsible ethics committee. Participation is voluntary, with written informed consent required. Data will be handled confidentially and analyzed in anonymized form only.

Risk-Benefit Assessment Risks are minimal and primarily related to routine blood draws (e.g., mild pain, bruising). Completing online questionnaires may cause fatigue or emotional discomfort; participants may pause or withdraw at any time.

Potential benefits include increased awareness of personal health progress and access to detailed feedback on biopsychosocial factors. Findings will contribute to improved, evidence-based psychosomatic care and support future research on integrative treatment models in Nutritional Psychiatry.

Dissemination of Results Findings from this pilot study will be disseminated through publication in peer-reviewed journals and presentations at scientific conferences. Authorship and publication will follow ICMJE guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

New patient at the outpatient clinic for Nutrition and Psychosomatics

Age between 18 and 65 years

Sufficient German language skills

Provided written informed consent

Able and willing to complete online questionnaires via email

Exclusion Criteria:

* Lack of consent or inability to provide informed consent

Diagnosed dementia (Mini-Mental State Exam < 20)

Severe substance dependence (e.g., alcohol, benzodiazepines, opioids)

Serious physical, neurological, or motor impairments preventing questionnaire completion

No access to or ability to use email for online forms

Diagnosis of cancer, severe autoimmune disease, or immunosuppression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress levels measured by the Perceived Stress Scale (PSS-10) | Baseline, 3 months, 6 months, 9 months, and 12 months
  The Perceived Stress Scale (PSS-10) is a validated 10-item self-report questionnaire that measures the degree to which situations in one's life are appraised as stressful. The scale assesses subjective stress over the past month. Scores range from 0 to 40, with higher scores indicating greater perceived stress. Changes in PSS-10 scores from baseline to 12 months will be analyzed to assess the effect of the nutrition-based care intervention on stress levels.

SECONDARY OUTCOMES:
Change in patient satisfaction | Baseline, 3 months, 6 months, 9 months, and 12 months
  Measured via a self-designed patient satisfaction questionnaire, covering areas such as care quality, communication, and organization
Brief Resilience Scale (BRS-D) Score | Baseline, 3 months, 6 months, 12 months
  The Brief Resilience Scale (BRS-D) assesses psychological resilience-specifically, the ability to bounce back from stress-through 6 items rated on a 5-point Likert scale.
  Unit of Measure: Units on a Scale Scale Range: 1 (low resilience) to 5 (high resilience) Interpretation: Higher scores indicate greater resilience (better outcome)
Somatic Symptom Scale (SSS-8) Score | Baseline, 3 months, 6 months, 12 months
  The Somatic Symptom Scale-8 measures the burden of physical symptoms using 8 items.
  Unit of Measure: Units on a Scale Scale Range: 0 (no symptoms) to 32 (very high symptom burden) Interpretation: Higher scores indicate greater physical symptom burden (worse outcome)
SF-12 Health Survey Score - Physical and Mental Components | Baseline, 3 months, 6 months, 12 months
  Description:
  The SF-12 assesses health-related quality of life via physical and mental health domains. Scores are standardized.
  Unit of Measure: Units on a Scale Scale Range: 0 (poor health) to 100 (excellent health) Interpretation: Higher scores indicate better physical or mental health (better outcome)
EQ-5D-5L Index Score | Baseline, 3 months, 6 months, 12 months
  The EQ-5D-5L evaluates five dimensions of health and provides a utility index score.
  Unit of Measure: Units on a Scale Scale Range: -0.281 (worst health state) to 1 (full health); country-specific Interpretation: Higher scores indicate better health-related quality of life (better outcome)
REAP-S v.2 Score (Rapid Eating Assessment - Short Version) | Baseline, 3 months, 6 months, 12 months
  The REAP-S v.2 is a brief dietary screener evaluating nutrition quality and eating patterns.
  Unit of Measure: Units on a Scale Scale: higher = healthier Interpretation: Higher scores generally reflect healthier dietary habits
OPD Score (Operationalized Psychodynamic Diagnostics) | Baseline, 6 months, 12 months
  The OPD instrument assesses psychodynamic functioning including interpersonal relations and internal conflicts.
  Unit of Measure: Units on a Scale Scale Range: Varies depending on subdomain (specify if available) Interpretation: Interpretation depends on axis; typically, higher dysfunction scores indicate worse outcome
Subjective Health Literacy | Baseline, 3 months, 6 months, 12 months
  ubjective health literacy is assessed by both participants and physicians using a 1-10 Likert scale at each time point.
Body Mass Index (BMI) [kg/m²] | Baseline, 3 months, 6 months, 9 months, and 12 months
  BMI will be calculated from measured height (in meters) and weight (in kilograms).
  Unit of Measure: kg/m² Scale Range: Typically 10-50 kg/m² Interpretation: Higher BMI indicates greater body mass; classified by WHO as underweight, normal, overweight, obese
Weight | Baseline, 3 months, 6 months, 9 months, and 12 months
  Body weight measured using a calibrated scale. Unit of Measure: kilograms Interpretation: Used to calculate BMI and assess weight changes
Height | Baseline, 3 months, 6 months, 9 months, and 12 months
  Height measured using a stadiometer. Unit of Measure: meters Scale Range: 1.3-2.2 m Interpretation: Used to calculate BMI
Differential Blood Count | Baseline, 3 months, 6 months, 9 months, and 12 months
  Complete blood count with differentiation (e.g., neutrophils, lymphocytes, eosinophils, monocytes, basophils).
  Unit of Measure: cells/µL or % Scale Range: Depends on cell type Interpretation: Reflects immune status and inflammation
C-Reactive Protein (CRP) | Baseline, 3 months, 6 months, 9 months, and 12 months
  CRP is a marker of systemic inflammation. Unit of Measure: mg/L Scale Range: <5 mg/L = normal Interpretation: Higher levels indicate acute or chronic inflammation
Interleukin-6 (IL-6) | Baseline, 3 months, 6 months, 9 months, and 12 months
  IL-6 is a pro-inflammatory cytokine. Unit of Measure: pg/mL Scale Range: <7 pg/mL normal (lab-specific) Interpretation: Elevated in systemic inflammation, infection, stress
Fasting Blood Glucose | Baseline, 3 months, 6 months, 9 months, and 12 months
  Measured after ≥8 hours of fasting. Unit of Measure: mg/dL Scale Range: 70-100 mg/dL Interpretation: Higher = impaired glucose metabolism or diabetes
HOMA-Index | Baseline, 3 months, 6 months, 9 months, and 12 months
  Homeostatic Model Assessment Index calculated from fasting glucose and insulin. Unit of Measure: Unitless Scale Range: ~0.5-2.5 normal Interpretation: Higher values suggest insulin resistance
Total Cholesterol | Baseline, 3 months, 6 months, 9 months, and 12 months
  Sum of HDL, LDL, and VLDL. Unit of Measure: mg/dL Scale Range: <200 mg/dL desirable Interpretation: Higher levels associated with cardiovascular risk
HDL Cholesterol | Baseline, 3 months, 6 months, 9 months, and 12 months
  High-density lipoprotein cholesterol - "good" cholesterol. Unit of Measure: mg/dL Scale Range: >40 (men), >50 (women) Interpretation: Higher values protective
LDL Cholesterol | Baseline, 3 months, 6 months, 9 months, and 12 months
  Low-density lipoprotein - "bad" cholesterol. Unit of Measure: mg/dL Scale Range: <130 mg/dL desirable Interpretation: Higher values increase atherogenic risk
Triglycerides | Baseline, 3 months, 6 months, 9 months, and 12 months
  Blood lipids, reflecting energy metabolism. Unit of Measure: mg/dL Scale Range: <150 mg/dL Interpretation: Higher = metabolic risk
Vitamin D (25-OH) | Baseline, 3 months, 6 months, 9 months, and 12 months
  Storage form of vitamin D Unit of Measure: ng/mL Scale Range: 20-50 optimal Interpretation: Low = deficiency; high = risk of toxicity
Ferritin | Baseline, 3 months, 6 months, 9 months, and 12 months
  Iron storage protein; also acute-phase reactant. Unit of Measure: ng/mL Scale Range: 20-300 ng/mL Interpretation: Low = iron deficiency, high = inflammation
Homocysteine | Baseline, 3 months, 6 months, 9 months, and 12 months
  Amino acid linked to B-vitamin status and cardiovascular risk. Unit of Measure: µmol/L Scale Range: <15 µmol/L Interpretation: Elevated = B12/B6/folate deficiency or oxidative stress
Vitamin B12 | Baseline, 3 months, 6 months, 9 months, and 12 months
  Water-soluble vitamin important for nerve and red blood cell function. Unit of Measure: pg/mL Scale Range: 200-900 pg/mL Interpretation: Low = deficiency with neuro/cognitive risks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Morkl S, Ramirez-Obermayer A, DelFabro B, Lackner S, Holasek S, Traub J, Grossbacher K, Brandstatter A, Wilding M, Wagner-Skacel J. Evaluation of the first nutritional psychiatry and psychosomatics outpatient clinic: Protocol for a prospective study of an individualized biopsychosocial therapy approach. PLoS One. 2026 Jan 5;21(1):e0339862. doi: 10.1371/journal.pone.0339862. eCollection 2026. PMID 41490357